CLINICAL TRIAL: NCT02996526
Title: The Incidence and Impact of Vocal Cord Dysfunction In Patients Undergoing Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Sadeesh Srinathan, MD, Dr. Sadeesh Srinathan Associate Professor Section of Thoracic Surgery, University of Manitoba
Other Study IDs: SSMGAD2016
Record Dates: First submitted 2016-08-19; First posted 2016-12-19 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Vocal Cord Paresis; Acquired Vocal Cord Palsy
Keywords: vocal cord palsy dysfunction thoracic surgery complication
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Intact Vocal Cord Mobility: Patients with normal laryngeal function post thoracic surgery
- Vocal Cord Dysfunction: Patients with abnormal vocal cord movement of 1 or both vocal cords post thoracic surgery

SUMMARY:
Population-based single centre, blinded, prospective cohort study of the impact of recurrent laryngeal nerve (RLN) injury on Thoracic Surgery patients. The principal outcome of interest is the effect of RLN injury on respiratory complications. Voice, swallowing, cardiac and mortality outcomes will also be determined.

DETAILED DESCRIPTION:
Objectives:

Primary: Estimate the prevalence of vocal cord dysfunction after thoracic surgery and the association of vocal cord dysfunction and immediate post operative respiratory complication after thoracic surgery.

Secondary:

1. Estimate the prevalence of vocal cord dysfunction in the pre-operative patient population undergoing thoracic surgery, i.e. the baseline prevalence.
2. Estimate the incidence of new vocal cord dysfunction in the post-operative period, i.e. the incidence of new dysfunction
3. Estimate the association of vocal cord dysfunction and respiratory, voice, swallowing, and mortality outcomes
4. Estimate the impact of vocal cord immobility on hospital length of stay, ICU admission rates and duration

Population: All patients undergoing thoracic surgery at Health Sciences Centre in Winnipeg, Canada. This is a tertiary care centre with a population-based referral base of 1.5 million people

Schematic of Study Design:

Enrollment Vocal Cord Mobility Assessment 1

Total N=141: Obtain informed consent. Screen potential participants by inclusion and exclusion criteria; obtain history Perform Flexible Nasolaryngoscopy by otolaryngology resident, document by videorecording

Vocal Cord Mobility Assessment 2 Post operative day 1-2 Perform Flexible Nasolaryngoscopy by otolaryngology resident, document by videorecording

Collection of functional outcomes Hospital Discharge or Death Collection of data on respiratory, voice, swallowing, cardiovascular mortality outcomes, hospital length of stay and ICU admission duration

Review of Vocal Cord Mobility Assessment by expert (Laryngologist) by review of videorecordings of nasolaryngoscopy

Statistical Analysis Final Assessments Association of vocal cord immobility and functional outcomes and death.

2.1 Background Information Research Question: In patients undergoing thoracic surgery, what is the incidence of respiratory and associated complications in the 30 day post-operative period among those with/without Recurrent Laryngeal Nerve (RLN) Injury?

Background: The issue of RLN injury is an important clinical challenge in thoracic surgery, as respiratory complications are the greatest source of morbidity in our surgical population . Clinical care experience and the literature demonstrate a high incidence of respiratory complications (20-60% incidence of pneumonia for esophagectomy and a 20% death rate for those who contract pneumonia) in the post-operative thoracic surgery population.

The thoracic surgery population is at uniquely elevated risk for respiratory complications due to the high prevalence of COPD, the nature of the primary surgical procedure directly diminishing pulmonary function and toilet; and possible RLN injury. The only modifiable element of this triad is RLN injury, and appears to be the most important element based on clinical experience and the limited literature available. The RLN supplies motor innervation to the vocal cords; vocal cord closure is considered the most important protective mechanism against aspiration into the lungs . Patients with a RLN injury demonstrate a 5-fold risk of contracting pneumonia, a 5-fold risk of reintubation or tracheostomy , and have 40-60% longer hospital stays than patients without RLN injury.

The current literature base is substantially lacking with regards to the incidence of RLN injury, with estimates varying from 4-80% based on retrospective reviews or prospective studies which fail to examine all patients. The highest quality studies demonstrate a RLN injury rate in the range of 20-40% for major procedures such as esophagectomy and pneumonectomy.

With the recent advent of injection laryngoplasty for vocal cord medialization, there is now a practical means of potentially altering the course of this pathologic triad. This procedure can be performed at the bedside under local anesthetic, allowing for early intervention in this high-risk population as a bulwark against aspiration.

Prospectively examining the incidence of pre and post-operative vocal cord immobility in all thoracic surgery patients is the only means to quantify the health burden associated with RLN injury.

Potential Risks Potential risks of the study include time involved in considering participation, providing consent and data such as subjective voice quality and undergoing flexible nasolaryngoscopy to assess vocal cord status. No health, economic or legal risks are anticipated for the participants.

Potential Benefits No direct benefit, either monetary or health improvement will accrue to patients from participation in the study.

Study Outcome Measures Vocal Cord Mobility - Flexible nasolaryngoscopy to visualize mobility status of vocal cords.

Voice - Voice Handicap Index 10. Validated instrument used for subjective assessment of voice, 10 plain language questions answered by the patient.

Respiratory: Incidence of pneumonia (as defined by CDC criteria) and intubation Swallowing: Oral diet vs NPO and diet texture tolerated at discharge Cardiovascular: Myocardial Infarction as defined by the third universal criteria 2012 by third ESC/ACCF/AHA/WHF, Cerebrovascular Accident as defined by WHO MONICA criteria and Neurology specialist consultation

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing thoracic surgery at Health Sciences Centre Winnipeg. Recruitment will be performed by the thoracic surgeon faculty within the Division of Thoracic Surgery. Written informed consent will be obtained from the patient by an independent research assistant.

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Provide signed and dated informed consent form.
* Willing to comply with all study procedures and be available for the duration of the study.
* Male or female, aged 18 and over..
* Have a condition requiring surgical entry into the thoracic cavity

Exclusion Criteria:

* All individuals meeting any of the exclusion criteria at baseline will be excluded from the study. Patients with severely deviated nasal anatomy precluding flexible nasolaryngoscopy Tracheostomy in situ Neurologic or developmental deficits impairing the ability to consent or cooperate with examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing thoracic surgery at Health Sciences Centre in Winnipeg, Canada. This is a tertiary care centre with a population-based referral base of 1.5 million people.
Sampling Method: Non-Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with vocal cord dysfunction assessed by nasolaryngoscopy on the first post-operative day | Post-operative day 1

SECONDARY OUTCOMES:
Number of patients with respiratory complictions | Within 30 days of operation
Number of patients with vocal cord dysfunction assessed by nasolaryngoscopy prior to operation | Day of operation
Hospital length of stay | From date of primary operation to discharge
  Number of days between admission to hospital and discharge
The number of patients with swallowing difficulties, cardiac complications and who have died | From the date of operation to day 30 after operation
ICU length of stay | From date of operation to discharge from hospital
  The total number of days admitted to the intensive care unit (a facility where full ventilator support and inotropic support can be provided) If more than one admission episode to the ICU, the total number of days in the ICU census is counted across the multiple admission episodes.
Readmission to hospital | From day of surgery to day 90 after operation
  Number of readmission episodes after initial discharge and during the 90 day period after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Sadeesh Srinathan, MD, Principal Investigator — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided